CLINICAL TRIAL: NCT01502306
Title: A Randomized Trial of Medi-Cal Beneficiaries Calling the California Smokers' Helpline
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); University of California, San Francisco (Other); California Department of Public Health (Other); California Department of Health Services (Other)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, Department of Family and Preventive Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMS NOA # 1B1CMS330882-01-00
Record Dates: First submitted 2011-12-23; First posted 2011-12-30 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Telephone; Self-help; Smoking abstinence; Incentives; Nicotine-replacement therapy; Medi-Cal; Medicaid
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telephone counseling (Experimental): One-on-one, proactive telephone counseling to quit smoking; The content of the counseling addresses both behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. Counseling begins immediately after intake, if the client is available for a 30-minute session or by appointment at the clients' convenience. Counseling includes a comprehensive pre-quit session (to include motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four proactive follow-up calls. The follow-up calls (about 10 minutes) will be scheduled as follows: a reminder call if the quit date is more than one week out for the initial counseling, on the quit date, 4-7 days after the quit date, and 10-14 days after the quit date.
  Interventions: Behavioral: Telephone counseling
- Phone counseling & nicotine patches (Experimental): One-on-one, proactive telephone counseling to quit smoking; The content of the counseling addresses both behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. Counseling includes a comprehensive pre-quit session (to include motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four proactive follow-up calls.
  Nicotine patches (four weeks' worth) are sent directly to clients the day after the screening intake. Dosage is 21 mg if smoking 11 or more per day, 14 mg if smoking 6-10 per day and 7mg if smoking <6 per day.
  Interventions: Drug: Nicotine patches
- Phone counseling, NRT and incentives (Experimental): One-on-one, proactive telephone counseling to quit smoking; The counseling addresses behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. Counseling includes a comprehensive pre-quit session (to include motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four proactive follow-up calls.
  Nicotine patches (four weeks' worth) are sent directly to clients. Dosage is 21 mg if smoking 11 or more per day, 14 mg if smoking 6-10 per day and 7mg if smoking <6 per day.
  Gift cards (to one of 4 major chains) are $20 for the first counseling session and $10 for each additional one (up to five sessions total).
  Interventions: Behavioral: Incentive

INTERVENTIONS:
Behavioral: Telephone counseling — Telephone counseling is conducted in the appropriate language (Spanish and English) by counselors at the California Smokers' Helpline. Counselors use a structured protocol and there is a record for each call. Quantitative information that will be available for analysis include: timing, length, and frequency of counseling calls.
  Arms: Telephone counseling
Drug: Nicotine patches — Clients will be screened for contraindications to nicotine patch use, and a doctor's approval will be necessary before patches are sent if a contraindication exists.
  Other Names: Habitrol
  Arms: Phone counseling & nicotine patches
Behavioral: Incentive — They will be given their choice of gift cards from one of 4 major business chains: Wal-Mart, Target, Vons/Safeway, or Ralph's/Kroger card.
  Arms: Phone counseling, NRT and incentives

SUMMARY:
California Smokers' Helpline will conduct a randomized trial to evaluate 3 strategies of services and/or incentives on smoking cessation rates. This project has the following specific aims:

1. To increase tobacco cessation among Medi-Cal beneficiaries who currently smoke, and to improve the management of diabetes and other chronic disease by means of tobacco cessation.
2. Demonstrate that tobacco cessation benefits that are well promoted and barrier free and include modest incentives, are effective in reducing smoking prevalence, lowering Medi-Cal health care costs, and improving health outcomes for diabetes management in particular.

DETAILED DESCRIPTION:
The mission of the California Department of Health Care Services (DHCS), California's single State Medicaid Agency, is to preserve and improve the health status of all Californians by operating and financing programs delivering effective health care services to eligible individuals. Medi-Cal (California's Medicaid Program) is the largest purchaser of health care in the state, serving over 7.5 million beneficiaries. Approximately half of all Medi-Cal beneficiaries receive their health care through managed care plans, while the other half receive care on a fee-for-service basis.

DHCS programs are designed to emphasize prevention-oriented health care measures (such as quitting smoking) that improve health and well-being, and ensure effective expenditure of public resources to serve those with the greatest health care needs. This study (MIPCD) aligns with the goals and objectives of the DHCS Strategic Plan, which states, "DHCS supports and values healthy lifestyle behaviors, and aims to promote the use of preventive, health improvement, and wellness services/activities."

The primary intervention in this study will be the internationally recognized, California Smokers' Helpline (Helpline) operated by the University of California, San Diego (UCSD). Established in 1992, more than 50% of the Helpline's clients are Medi-Cal members. In this study, the Helpline will: operate a fully functioning quitline call center with trained personnel and live capabilities in English, Spanish, Mandarin, Cantonese, Korean and Vietnamese; assess eligibility for the randomized trial; obtain consent for participation in the trial; send individually tailored self-help materials to registered participants; provide one-on-one telephone counseling, including a comprehensive, pre-quit planning session and up to four relapse-prevention sessions; evaluate the services provided; maintain detailed, confidential records of each beneficiary's cessation activity and receipt of incentives and services. Callers with a valid Medi-Cal ID who have diabetes or other eligible condition(s) and provide consent for the study will be randomized into one of the three arms of the trial. The arms of the trial are detailed below:

1. Group 1 (Policy A) - current policy: beneficiaries who call the Helpline will get free counseling and a certificate of enrollment, which is required in order for them to obtain free nicotine replacement therapy (NRT) from their pharmacy, four weeks' worth at a time. Beneficiaries can receive two courses of treatment per year.
2. Group 2 (Policy B1) - a new policy in which beneficiaries who call the Helpline get free counseling and have free nicotine patches shipped directly to their home, with no limit on the number of quit attempts they can make in a year.
3. Group 3 (Policy B2) - a variant of B1 in which beneficiaries will get free counseling and free nicotine patches shipped directly to their home, with no annual limit on quit attempts. Participants will also get an added incentive to adhere to the counseling program, in the form of gift cards worth $20 for their initial counseling call and $10 for each additional follow-up counseling call (up to five sessions total, or $60).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Medi-Cal beneficiary with valid Medi-Cal beneficiary ID
* Willing to link Helpline data with Medi-Cal utilization data
* English or Spanish speaking
* Valid phone number
* Valid address
* Gave consent to participate in study and evaluation

Exclusion Criteria:

* Contraindication(s) to nicotine patches and no MD approval
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3816 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego; California Smokers' Helpline, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu SH, Stretch V, Balabanis M, Rosbrook B, Sadler G, Pierce JP. Telephone counseling for smoking cessation: effects of single-session and multiple-session interventions. J Consult Clin Psychol. 1996 Feb;64(1):202-11. doi: 10.1037//0022-006x.64.1.202. PMID 8907100
- [Background] Zhu SH, Anderson CM, Tedeschi GJ, Rosbrook B, Johnson CE, Byrd M, Gutierrez-Terrell E. Evidence of real-world effectiveness of a telephone quitline for smokers. N Engl J Med. 2002 Oct 3;347(14):1087-93. doi: 10.1056/NEJMsa020660. PMID 12362011
- [Background] Anderson CM, Zhu SH. Tobacco quitlines: looking back and looking ahead. Tob Control. 2007 Dec;16 Suppl 1(Suppl 1):i81-6. doi: 10.1136/tc.2007.020701. PMID 18048638
- [Background] Lynagh MC, Sanson-Fisher RW, Bonevski B. What's good for the goose is good for the gander. Guiding principles for the use of financial incentives in health behaviour change. Int J Behav Med. 2013 Mar;20(1):114-20. doi: 10.1007/s12529-011-9202-5. PMID 22094998
- [Derived] Anderson CM, Cummins SE, Kohatsu ND, Gamst AC, Zhu SH. Incentives and Patches for Medicaid Smokers: An RCT. Am J Prev Med. 2018 Dec;55(6 Suppl 2):S138-S147. doi: 10.1016/j.amepre.2018.07.015. PMID 30454668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was between July 2012 and May 2013
Groups:
- Phone Counseling & Nicotine Patches: One-on-one, proactive telephone counseling to quit smoking; The content of the counseling addresses both behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. Counseling includes a comprehensive pre-quit session (to include motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four proactive follow-up calls.
  Nicotine patches (four weeks' worth) are sent directly to clients the day after the screening intake. Dosage is 21 mg if smoking 11 or more per day, 14 mg if smoking 6-10 per day and 7mg if smoking <6 per day.
  Nicotine patches: Clients will be screened for contraindications to nicotine patch use, and a doctor's approval will be necessary before patches are sent if a contraindication exists.
- Phone Counseling, NRT and Incentives: One-on-one, proactive telephone counseling to quit smoking; The counseling addresses behavioral and cognitive issues that the individual smoker faces in his/her attempt to quit. Counseling includes a comprehensive pre-quit session (to include motivation, planning, setting of a quit date and the discussion of quitting aids including nicotine patch use) plus up to four proactive follow-up calls.
  Nicotine patches (four weeks' worth) are sent directly to clients. Dosage is 21 mg if smoking 11 or more per day, 14 mg if smoking 6-10 per day and 7mg if smoking <6 per day.
  Gift cards (to one of 4 major chains) are $20 for the first counseling session and $10 for each additional one (up to five sessions total).
  Incentive: They will be given their choice of gift cards from one of 4 major business chains: Wal-Mart, Target, Vons/Safeway, or Ralph's/Kroger card.
Period: Overall Study
Arm/Group | Telephone Counseling | Phone Counseling & Nicotine Patches | Phone Counseling, NRT and Incentives
Started | 1004 | 1405 | 1407
Completed | 1004 | 1405 | 1407
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Counseling | Phone Counseling & Nicotine Patches | Phone Counseling, NRT and Incentives | Total
Number analyzed (Participants) | 1004 | 1405 | 1407 | 3816
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 53 | 67 | 63 | 183
  25-44 | 355 | 515 | 499 | 1369
  45-64 | 550 | 743 | 761 | 2054
  >=65 | 46 | 80 | 84 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 675 | 955 | 953 | 2583
  Male | 329 | 450 | 454 | 1233
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 616 | 819 | 819 | 2254
  Black | 159 | 275 | 283 | 717
  Hispanic | 91 | 142 | 138 | 371
  Asian/Pacific Islander | 19 | 24 | 16 | 59
  American Indian | 19 | 38 | 31 | 88
  Multi-Racial | 99 | 103 | 114 | 316
  Other | 1 | 4 | 6 | 11
Education [Count of Participants; unit: Participants]
  <= 12 | 590 | 844 | 823 | 2257
  >12 | 414 | 561 | 584 | 1559

OUTCOME MEASURES:

1. Primary Outcome: 30-day Abstinence
Description: At a given point in time (in this case, 7 months after program registration), quitline participants are asked whether they have used cigarettes or other forms of tobacco in the past 30 days. Those who reply that they have not used tobacco in the past 30 days are considered to have quit.
Time Frame: 7 months post enrollment
Population: Number of participants analyzed reflects the number of participants the quitline was able to reach at 7-months
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Counseling | Phone Counseling & Nicotine Patches | Phone Counseling, NRT and Incentives
Number analyzed (Participants) | 639 | 919 | 958
Participants | 168 | 237 | 302

2. Secondary Outcome: Percentage of Smokers Making a 24-hour Quit Attempt
Description: At a given point in time (in this case, 2 months after program registration), quitline participants are asked whether they made a quit attempt (attempt at quitting smoking) and how long they made it.
Time Frame: 2 months post enrollment
Population: Number of participants analyzed reflects the number of participants the quitline was able to reach at 2-months
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Counseling | Phone Counseling & Nicotine Patches | Phone Counseling, NRT and Incentives
Number analyzed (Participants) | 789 | 1093 | 1143
Participants | 546 | 847 | 962

3. Secondary Outcome: Continuous Abstinence Rates for Those Who Made Quit Attempts
Description: Not smoking since the quit date
Time Frame: 7-months post enrollment
Population: Number of participants analyzed reflects the number of participants the quitline was able to reach at 7-months
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Counseling | Phone Counseling & Nicotine Patches | Phone Counseling, NRT and Incentives
Number analyzed (Participants) | 639 | 919 | 958
Participants | 90 | 145 | 185

4. Secondary Outcome: 7-day Prevalence.
Description: Seven-day point prevalence abstinence is a measure of, in this case, tobacco cessation outcomes for quitlines. At a given point in time (in this case, 7 months after program registration), quitline participants are asked whether they have used cigarettes or other forms of tobacco in the past 7 days.
Time Frame: 7-months post enrollment
Population: Number of participants analyzed reflects the number of participants the quitline was able to reach at 7-months
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Counseling | Phone Counseling & Nicotine Patches | Phone Counseling, NRT and Incentives
Number analyzed (Participants) | 639 | 919 | 958
Participants | 162 | 231 | 298

ADVERSE EVENTS:
Arm/Group | Telephone Counseling | Phone Counseling & Nicotine Patches | Phone Counseling, NRT and Incentives
Serious Adverse Events (participants affected / at risk) | 0/1004 | 0/1405 | 0/1407
Other Adverse Events (participants affected / at risk) | 0/1004 | 0/1405 | 0/1407

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No